CLINICAL TRIAL: NCT04159129
Title: Effects of a Three-week Inpatient Pulmonary Rehabilitation Program on Walking Speed in Patients With Chronic Obstructive Pulmonary Disease (COPD) or Interstitial Lung Diseases (ILD)
Brief Title: Effects of Pulmonary Rehabilitation on Walking Speed in Patients With COPD or ILD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: Psychologische Hochschule Berlin (Unknown)
Responsible Party: Principal Investigator, Klaus Kenn, Prof. Dr. Klaus Kenn, Schön Klinik Berchtesgadener Land
Other Study IDs: Ampel2019
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial
Keywords: walking speed; dyspnoe; stress; anxiety; traffic light
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the effects of a three-week inpatient pulmonary rehabilitation (PR) program on the walking speed in patients with chronic obstructive (COPD) or interstitial lung disease (ILD).

DETAILED DESCRIPTION:
At most german traffic light crossings, a walking speed of 1,2m/sec is required to cross the road in time. Patients who are unable to cross the road at this speed, expose themselves to an increased level of stress and possibly the risk of accidents. Thus, they are discouraged from participating in an active social life.

An UK study (Nolan et al., Thorax 2018) showed that only 10.7% of the 926 patients with moderate COPD attained a walking speed of 1.2m/sec. As PR plays a key role in the management of chronic lung diseases in order to improve patients´ exercise capacity, the aim of this study was to evaluate the PR effects on the Walking Speed in patients with COPD or ILD. The investigators hypothesize that PR improves the ability to cross the road in the appropriate time.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a pulmonary Rehabilitation program (Schön Klinik BGL)
* Indication: COPD or ILD
* COPD; FEV1 <50%
* ILD: FVC <70%
* written informed consent

Exclusion Criteria:

* non compliance

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with COPD or ILD who fulfill the inclusion criteria will be recruited during an inpatient pulmonary Rehabilitation program.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
change of maximum walking speed | Day 1 and Day 21
  assessed during a walk of 11m

SECONDARY OUTCOMES:
Change of usual walking Speed | Day 1 and Day 21
  assessed during a walk of 11m by using the individual daily life Walking Speed.
Change in balance | Day 1 and Day 21
  measured by the Leonardo platform
Change in walking speed during a field walk test | Day 1 and Day 21
  measured by the time needed to cross a traffic light (distance: 11m)
Change in tension symptoms during a field walk test | Day 1 and Day 21
  intensity of perceived tension symptoms experienced when crossing a traffic light (VAS scale, ranging from 0 to 10)
Change of exercise capacity | Day 1 and Day 21
  measured by the sit-to-stand test, test duration: 1 minute
Change in maximum leg strength | Day 1 and Day 21
  measured by the microfet, knee Extension
Change in anxiety and Depression symptoms | Day 1 and Day 21
  Anxiety/Depression measured by Hospital Anxiety and Depression Scale (HADS) - a screening questionnaire including seven questions each about Depression and Anxiety; each part ranging from 0 to 21; higher scores indicate higher presence of the respective state
Change of frailty (FFP) | Day 1 and Day 21
  measured by Fried Frailty Phenotype (FFP), including five constructs (weight loss, exhaustion, physical activity, gait speed and weakness); range 0-5, higher scores reflect increased Frailty: A score of 0 is considered as "robust", a score of 1-2 is considered as "pre-frail", a score lower than 2 reflects "Frailty"
Change in Quality of life: Chronic Respiratory Disease Questionnaire (CRQ) | Day 1 and Day 21
  assessed by the Chronic Respiratory Disease Questionnaire (CRQ)- a 20-item self-report questionnaire; score 1-7; higher scores indicate a better health-related quality of life
Change in illness perception | Day 1 and Day 21
  assessed by the Illness perception Questionnaire, revised (IPQ-R) - 18 items, score 1-5; higher scores indicate a worse illness perception, except of item 7,9,10,11,12.
Change in COPD-related fears on disease-specific disability | Day 1 and Day 21
  assessed by the German "COPD Angst Fragebogen" (CAF) - a 20-item self-report questionnaire, rated on a Lickert-scale (score 0-4); highest maximum score: 80 points; higher scores indicate higher anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof., Principal Investigator — Schön Klinik Berchtesgadener Land
Locations (1):
- Schön Klinikum Berchtesgadener Land, Schönau am Königssee, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No